CLINICAL TRIAL: NCT06553248
Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of GZR4 in Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GZR4 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GZR-CH1016
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Diabetes
Keywords: GZR4; PK; PD
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR4 (Experimental): s.c., once weekly
  Interventions: Drug: GZR4
- Insulin Degludec (Active Comparator): s.c., once daily
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: GZR4 — Administered once weekly subcutaneously (s.c., under the skin) for 6 weeks
  Arms: GZR4
Drug: Insulin Degludec — Administered once daily subcutaneously (s.c., under the skin) for 6 weeks
  Arms: Insulin Degludec

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of mutiple-dose GZR4 in subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female at the age of 18-65 (inclusive) at the time of informed consent
* Body mass index (BMI) between 18.5 and 35 kg/m2 (inclusive) at screening
* Diagnosis of type 2 diabetes mellitus for over 3 months
* Hemoglobin A1c (HbA1c) ≥ 6.5% and ≤ 10.0% at screening.

Exclusion Criteria:

* History of drug abuse within 1 year before screening, or positive drug abuse screening results during the screening period or at baseline
* Malignancy or increased risk of malignancy before screening: any suspected and/or diagnosed malignancy or documented history of malignancy
* Confirmed or suspected type 1 diabetes mellitus, gestational diabetes mellitus, or specific types of diabetes mellitus from other causes (monogenic diabetes syndrome, cystic fibrosis, pancreatitis, drug-induced or chemically induced diabetes mellitus, etc.) prior to screening
* Presence of the following diseases within 6 months prior to screening: diabetic ketoacidosis, diabetic lactic acidosis, or hyperosmolar nonketotic diabetic coma; proliferative retinopathy or maculopathy that is unstable or requiring treatment; symptomatic diabetic neuropathy, intermittent claudication or diabetic foot
* Severe hypoglycaemic events (Level 3 hypoglycaemia) within 6 months prior to screening, or 3 or more hypoglycaemic events (blood glucose ≤ 3.9 mmol/L) within 1 month prior to screening, or recurrent hypoglycaemia-related symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAE | Baseline to Week 6

SECONDARY OUTCOMES:
AUC0-inf | Week 6
AUC0-last | Week 6
AUC0-168h | Week 1, Week 6
Tmax,GZR4 | Week 1, Week 6
ADA of GZR4 | Baseline to Week 10

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No